CLINICAL TRIAL: NCT05046561
Title: Study to Reinforce Immunity (STRI) - A Phase 2 Double-Blind, Randomized, Placebo-Controlled Study to Investigate The Safety and Efficacy of STRI Formula in Non-Hospitalized Participants With COVID-19
Brief Title: Study to Reinforce Immunity (STRI) Phase 2 Clinical Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eyecheck, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: STRI12
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Covid19
Keywords: Covid-19 symptoms
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STRI Formula (Active Comparator): STRI Formula 3 capsules by mouth twice daily for 10 days
  Interventions: Drug: STRI Formula
- Placebo (Placebo Comparator): Placebo 3 capsules by mouth twice daily for 10 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STRI Formula — STRI Formula is a combination of food based substances (botanicals, vitamins, minerals, and protein) with multiple, distinct, synergistic, direct and indirect antiviral effects against SARS-CoV-2
  Arms: STRI Formula
Drug: Placebo — Placebo oral capsule
  Arms: Placebo

SUMMARY:
Protocol STRI12 - Study to Reinforce Immunity (STRI) - A Phase 2 Double-Blind, Randomized, Placebo-Controlled Study to Investigate the Safety and Efficacy of STRI Formula in Non-Hospitalized Participants with COVID-19 (the Study)

DETAILED DESCRIPTION:
The Study to Reinforce Immunity (STRI) Phase 2 Clinical Trial is a randomized, double-blind, placebo-controlled clinical trial protocol assessing the safety and efficacy of STRI Formula in non-hospitalized participants with COVID-19. STRI Formula is a combination of food-based substances designed specifically to combat SARS-CoV-2, the coronavirus that causes COVID-19.

The primary objective of the Study is to assess the efficacy of STRI Formula in reduction of time from treatment initiation to initial meaningful clinical improvement in COVID-19 symptoms. Additional secondary objectives are as follows:

1. To assess the safety of STRI Formula
2. To assess the efficacy of STRI Formula in reduction of time to COVID-19 sustained symptom improvement
3. To assess the efficacy of STRI Formula in reduction of time to COVID-19 initial symptom resolution
4. To assess the efficacy of STRI Formula in reduction of time to COVID-19 sustained symptom resolution
5. To assess the efficacy of STRI Formula in reduction in need for hospitalization
6. To assess the efficacy of STRI Formula in reduction in rates of fever
7. To assess the efficacy of STRI Formula in reduction in rates of hypoxia

ELIGIBILITY:
Inclusion Criteria:

1. Adults residing in the United States aged 18 years or older.
2. Provision of documentation of positive SARS-CoV-2 testing (via RT-PCR, rapid antigen testing) performed less than 7 days before screening, either via direct upload or confirmation from PCP.

   1. electronic secure document upload;
   2. allowing STRI Personnel to contact the PCP to confirm diagnosis; or
   3. allowing STRI Personnel to contact the laboratory where the RT-PCR analysis was performed
3. Initial date of onset of COVID-19 signs/symptoms 7 days or less from date of STRI Screening and Randomization (i.e., Day 0).
4. During screening (Day 0):

   1. participant-reported response of "Mild" or "Moderate" in response to the question "Overall, how severe were your infection symptoms today?" (FLU-PRO Plus Global Additional Daily Diary Items Question 1)
   2. During prescreening, participant self-reported response of "A little worse" or "Somewhat worse" or "Much worse" or "About the same" in response to the question "Overall, how were your infection symptoms today compared to yesterday?" (FLU-PRO Plus Global Additional Daily Diary Items Question 2)
   3. During prescreening, participant-reported response of "No" in response to the question "Have you returned to your usual health today?" (FLU-PRO Plus Global Additional Daily Diary Items Question 6)
   4. At least TWO participant self-reported responses of "Somewhat," "Quite A Bit," or "Very Much" in any FLU-PRO Plus domain other than smell and taste (i.e., nose, throat, eyes, chest/respiratory, head, gastrointestinal, or body/systemic domains)
5. Ability to self-measure and self-report body temperature, and peripheral oxygen saturation (with STRI provided thermometer and STRI provided pulse oximeter).
6. Provision of signed and dated electronic informed consent form (via 21 CFR Part 11 compliant platform).
7. Provision of participant's primary care physician (PCP) name and phone number.
8. Consent to allow STRI Personnel to contact PCP for any reason and discuss participant's medical history and/or obtain participant's medical records.
9. Stated willingness to comply with all study procedures and availability for the duration of the study, including intent to comply with lifestyle considerations throughout Study duration.
10. Ability to take oral medication and be willing to adhere to the STRI Intervention Product (STRI Formula or placebo as capsules) regimen.
11. Ability to use the internet daily and check email daily.
12. Ability and consent to send and receive SMS text messages via cellular phone.
13. Provision of information (name, email address, and cellular phone number) of an emergency contact (e.g., family member/friend/colleague) willing to communicate with STRI Personnel in case the participant deteriorates.
14. Willingness to discontinue any dietary supplement that contains any active ingredient in STRI Formula (ascorbic acid, cholecalciferol, zinc, copper, quercetin, hesperidin, caffeic acid, epigallocatechin gallate, bovine lactoferrin) for the duration of the Study.
15. For men and women with child-bearing potential (as defined below), willingness to use adequate contraception for at least 100 days after beginning the Study.

Exclusion Criteria:

1. Inability to comply with study or follow-up procedures, or provide regular updates to their health status when contacted by the STRI Personnel via email, SMS, or phone.
2. Any prior or current hospitalization for COVID-19 or any need for hospitalization for any reason.
3. Any prior or current treatment with any agent for COVID-19.
4. Any known allergies or known toxicities to any of the specific ingredients in STRI Formula (including ascorbic acid, vitamin D, zinc, copper, amla, caffeic acid, coffee, bovine lactoferrin, milk, quercetin, hesperidin, oranges, citrus fruits, and/or green tea)
5. Body Mass Index > 40 based on participant-reported weight and participant-reported height.
6. Participant-reported weight of less than 35kg.
7. Any history of radiation or chemotherapy for cancer within the last 3 months.
8. Any history of cardiac arrythmias, hemochromatosis, renal (including any known GFR < 60mL/min) or hepatic disease (including chronic liver disease).
9. Any history of chronic pulmonary disorders
10. Any history of any gastrointestinal surgery or disease (including bariatric surgery or gastrointestinal resection, inflammatory bowel disease, or chronic intestinal diseases, such as (but not limited to) eosinophilic enteritis or autoimmune enteritis).
11. Any history of mineral or vitamin overload or deficiency (including chronic iron overload states, copper overload states, or ascorbic acid, vitamin D, zinc, or copper deficiencies).
12. Any history of any adverse event to green tea extract or any herbal products.
13. Prescreening Alcohol Use Disorders Identification Test (AUDIT) score of 8 or more indicating hazardous or harmful alcohol consumption, or alcohol dependence.
14. Pregnant or nursing/breastfeeding participants or participants intending to become pregnant within the next 24 months.
15. Men or premenopausal women not using adequate contraception.
16. Any other factors as judged by the principal investigator that would cause harm or increased risk to the participant or preclude the participant's full adherence with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 598 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Length of time from treatment initiation to initial meaningful clinical improvement as measured over 30 days. | 30 days

SECONDARY OUTCOMES:
Proportion of participants with any recorded serious adverse events | 30 days
Proportion of participants with any new comprehensive metabolic panel abnormalities (including electrolyte levels, glucose levels, renal and liver function testing) related to STRI Intervention Product between baseline and 30 days. | 30 days
Proportion of participants with any new complete blood count abnormalities (including white blood cell, red blood cell, hemoglobin, and platelets) related to STRI Intervention Product between baseline and 30 days. | 30 days
Proportion of participants that develop fever (measured as body temperature of more than 100.4 degrees F using a participant self-recorded thermometer). | 30 days
Proportion of participants that develop hypoxia (measured as peripheral oxygen saturation of less than 93% using a participant self-recorded pulse oximeter). | 30 days
Length of time from treatment initiation to sustained meaningful clinical improvement. | 30 days
Length of time from treatment initiation to initial clinical recovery. | 30 days
Length of time from treatment initiation to sustained clinical recovery. | 30 days
Proportion of participants requiring hospitalization. | 30 days
Proportion of participants with COVID-19 signs/symptoms. | 30 days
Proportion of participants with COVID-19 signs/symptoms | 60 days
Proportion of participants who have expired. | 30 days
Proportion of participants who have expired. | 60 days

OTHER OUTCOMES:
Proportion of participants with PCR positivity for SARS-CoV-2 at 5, 10, 15, and 30 in saliva samples (first-stage only) compared to Day 1 (before treatment initiation) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rama D Jager, MD, Principal Investigator — Eyecheck, Inc.
Locations (13):
- United States (13):
  - Luna Research, Coral Gables, Florida
  - Prohealth Research Center, Doral, Florida
  - Solution Clinical Research, Doral, Florida
  - South Florida Research, Medley, Florida
  - G+C Research Group, Miami, Florida
  - Dynamic Medical Research, Miami, Florida
  - Vista Health, Miami, Florida
  - Davila Medical Research, Miami, Florida
  - A&A Research Group, Miami, Florida
  - The Miami Research Group, Miami, Florida
  - Affinity Clinical Research, Tampa, Florida
  - Beat COVID, Oak Forest, Illinois
  - Dorisca Research Consulting, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed, the de-identified, archived data may be transmitted to and stored for use by other researchers including those outside of the study. Permission to transmit de-identified data to other researchers has been included in the informed consent.
  Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint by contacting the PI.
Supporting Information: CSR
Time Frame: Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint by contacting the PI.
Access Criteria: Users of the STRI Dataset will be required to agree to terms that prohibit unlawful uses and intentional violations of privacy and require attribution.